CLINICAL TRIAL: NCT03370822
Title: A Mixed Methods Study to Explore the Feasibility of a Novel Continuous Fetal Monitoring
Brief Title: A Mixed Methods Study to Explore the Feasibility of a Novel Continuous Fetal Monitoring Device
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Other Study IDs: 201920
Record Dates: First submitted 2017-11-24; First posted 2017-12-12 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Fetal Distress; Fetal Heart Rate Disorder Nos
Keywords: Fetal monitoring; Acceptability; Fetal Heart Rate
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Women who have continuous fetal monitoring using the MONICA AN24 device. The MONICA AN24 is a wearable monitor with five adhesive electrodes placed on the mother's abdomen. This records the fetal heart rate, maternal heart rate and uterine contractions.
  Interventions: Device: MONICA AN24 device

INTERVENTIONS:
Device: MONICA AN24 device — Application of MONICA AN24 device and recording for the longest period of fetal heart rate recording possible (limited by battery life)

SUMMARY:
A stillbirth describes when a baby dies after 24 weeks of pregnancy and before being born. In the UK there are roughly 9 stillbirths every day. Normally, before a stillbirth occurs changes such as a slower heart rate and reduced movement take place. Fetal monitoring attempts to detect these changes so that babies can be delivered before they become severely ill. If a baby could be monitored continuously then these changes could be detected earlier. However, current forms of fetal monitoring, such as ultrasound, cannot be used for long periods of time and do not significantly reduce stillbirth rates. The Monica AN24 device is a continuous monitor which records the baby's heart rhythm using sensors placed on the mother's abdomen. As this is a new device there is little evidence about how well it works. In this project women will be asked how they feel about the device after wearing it. Doctors and midwives will also be asked about their views of the device. The effect of the mother's movement and the age of the baby on how well the Monica AN24 can record the baby's heart rhythm will also be assessed.

DETAILED DESCRIPTION:
In the United Kingdom (UK) stillbirth is defined as the death of a fetus before birth and after 24 weeks gestation. The incidence of stillbirth in the UK was 4.6 per 1000 in 2014. The annual rate of reduction was 1.4%, a rate considerably lower than other high income countries, such as Poland (4.5%) and Netherlands (6.8%), demonstrating that more can be done to reduce stillbirth rates in the UK. Stillbirths are often preceded by a series of adaptive changes, including changes in fetal heart rate (FHR) and reduced fetal movement. Fetal monitoring serves, in part, to identify these changes so that appropriate intervention can be initiated and adverse outcomes prevented. However, currently used forms of fetal monitoring, including Doppler ultrasound and cardiotocography, cannot provide an objective, longitudinal view of fetal wellbeing and do not significantly reduce stillbirth rates. A continuous fetal monitor could identify signs of fetal compromise earlier.

A recent study found that 45.1% of surveyed clinicians thought that a continuous fetal monitor would be beneficial to their practice, although 81.7% also expressed concerns about the utility and clinical implementation of such a device. The Monica AN24 monitor is a novel continuous fetal monitoring device which records the fetal electrocardiogram (fECG) via trans-abdominal electrodes. Monica AN24 has been shown to have good recording quality though one study reported an association between recording quality and gestational age. The effect of the device on maternal anxiety is not known. All studies assessing acceptability of the device to women have focused on the intrapartum period or during induction of labor. Consequently, a prospective observational cohort study is needed to assess the acceptability of the Monica AN24 device in the context of antenatal care, as is further exploration of factors affecting recording quality of the Monica AN24 device.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies attending St. Mary's Hospital, Manchester for antenatal care
* No abnormality identified on ultrasound scan of fetal biometry and umbilical and fetal Doppler indices
* Gestational age >24 weeks
* Able to give informed consent

Exclusion Criteria:

* Multiple pregnancies
* Maternal age <18 years
* Individuals who do cannot speak or do not understand fluent English
* Individuals unable to give informed consent
* Women in active labour

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Women who have an uncomplicated pregnancy attending the Research Clinics at St Mary's Hospital, Manchester.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Mother's experience of wearing device | Immediately following the period (usually 12-24 hours) of wearing MONICA AN24 device
  Qualitative Interview conducted within 24 hours of wearing the AN24 device
Change in Maternal Anxiety (GAD-2) | Maternal completion of the GAD-2 questionnaire before wearing the MONICA AN24 device and immediately following the period of wearing the MONICA AN24 device.
  Change in maternal anxiety as assessed by Generalised Anxiety Disorder 2 item (GAD-2)
Change in Maternal Anxiety (Pregnancy Specific Anxiety Score) | Maternal completion of the Pregnancy Specific Anxiety Score questionnaire before wearing the MONICA AN24 device and immediately following the period of wearing the MONICA AN24 device.
  Change in maternal anxiety as assessed by Pregnancy Specific Anxiety Score
Maternal Anxiety (STAI) | Maternal completion of the STAI before wearing the MONICA AN24 device and immediately following the period of wearing the MONICA AN24 device.
  Change in maternal anxiety as assessed by State Trait Anxiety Index.

SECONDARY OUTCOMES:
Recording quality - defined as the percentage of time the device recorded the fetal heart rate | During the 12-24 hour recording period
  The recording quality of the Monica AN24 device defined as the percentage of time the device recorded the fetal heart rate) with differing levels of maternal activity and differing gestational ages.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No